CLINICAL TRIAL: NCT05894187
Title: Exploring the Effects of an Informative Animated Video on Preoperative Anxiety in Children Undergoing Elective Otoplasty and Their Parents
Brief Title: The Impact of an Animated Video on Preoperative Anxiety in Children Undergoing Elective Otoplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Michael Bezuhly, Head, Division of Plastic & Reconstructive Surgery Director, Craniofacial Program IWK Health Centre, IWK Health Centre
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1028283
Record Dates: First submitted 2023-05-21; First posted 2023-06-08 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Pre-operative Anxiety; Otoplasty; Paediatric Surgery
Keywords: otoplasty; pre-operative anxiety; animated video

STUDY DESIGN:
Intervention Model Description: prospective, randomized, single-blind controlled superiority
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (no video) (No Intervention): Children in this group will not receive a link to view an informational animated prior to their surgery date
- Intervention group ( video) (Experimental): Children in this group will receive a link to view an informational animated video 3 nights prior to their surgery date.
  Interventions: Other: animated video

INTERVENTIONS:
Other: animated video — Participants randomized to the intervention group will receive a link to a short survey gauging parent anxiety levels three days prior to their childs surgery date. If randomly assigned to watch the informative animated video, the survey will be followed by a link to a video which families are free to watch prior to your child's surgery date. Once participants and there family watch the video, they will be asked to rate the quality of the video on a scale of 0 (very bad) to 10 (excellent). Responses to this question will be used to confirm that participants watched the video to the end.
  Arms: Intervention group ( video)

SUMMARY:
The study is a prospective, randomized, single-blind controlled superiority trial to evaluate the effect of viewing an informative animated video a day prior to surgery on preoperative anxiety in pediatric patients scheduled for elective otoplasty. The primary outcome will be modified Yale Preoperative Anxiety Scale (mYPAS) score at the time of general anesthesia induction compared between families that were assigned to view the animated video the day before and those that were not. The participants for this study will be children undergoing elective otoplasty at the IWK Health Centre. Those participants randomized to the intervention group will receive a link to a short survey gauging parent anxiety levels. The survey will be followed by a link to an informative animated video which the participants and their families will watch. The control group will be participants assigned not to receive the email link to the informative animated video.

ELIGIBILITY:
Inclusion Criteria:

* They are undergoing an otoplasty alone with no other procedures on the same day
* The patient must not have previously undergone an otoplasty; the patient must be between the ages of 4 and 12;
* The patient must understand spoken English;
* The participating parent must be able to read English at a grade six level; and the patient should not have received premedication.

Exclusion Criteria:

* Under the age of 4 or over the age of 12
* Have not undergone a previous otoplasty

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
modified Yale Preoperative Anxiety Scale (mYPAS) | Data acquisition will occur within 24 hours. Recording will start once patient enters room and is positioned on OR table. Recording will stop one minute after induction mask is put on patient. Total recording time will be five minutes.
  The mYPAS is a validated observational measure to assess the behaviour of children of all ages preoperatively and consists of 27 items divided into five domains (activity, emotional status, arousal state, vocalization, and use of parents).24,27,28 The mYPAS scores range from 22 to 100, with higher values indicating greater anxiety. The mYPAS is considered the gold-standard for observational preoperative anxiety assessment in paediatric patients.24,27-30

SECONDARY OUTCOMES:
parental self-reported anxiety using the State-Trait Anxiety Inventory | Within 48 hours prior to arrival at the IWK for surgery and again upon arrival at the IWK immediately prior to their child leaving the waiting area to enter the operating room
  The STAI, which consists of two 20-item subscales measures is self-administered on a four-point scale for each item. The scores for each of the subscales range from a minimum of 20 to a maximum of 80, the higher scores suggest the greater psychological anxiety. The tool was designed to differentiate between the temporary condition of "state anxiety" in response to an acute event and the more general and long-standing quality of "trait anxiety" entrenched in the individual's personality. This tool has been validated in a variety of clinical settings including parental anxiety prior to a child's surgery.26
modified Yale Preoperative Anxiety Scale (mYPAS) | mYPAS score while in the preoperative waiting area
  The mYPAS is a validated observational measure to assess the behaviour of children of all ages preoperatively and consists of 27 items divided into five domains (activity, emotional status, arousal state, vocalization, and use of parents).24,27,28 The mYPAS scores range from 22 to 100, with higher values indicating greater anxiety. The mYPAS is considered the gold-standard for observational preoperative anxiety assessment in paediatric patients.24,27-30

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bezuhly, MD, Principal Investigator — IWK Health Centre
Locations (1):
- IWK health centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Spielberger CD. Manual for the State-Trait Anxiety Inventory. Palo Alto: Consulting Psychologists Press, 1983.
- [Background] Heeren A, Bernstein EE, McNally RJ. Deconstructing trait anxiety: a network perspective. Anxiety Stress Coping. 2018 May;31(3):262-276. doi: 10.1080/10615806.2018.1439263. Epub 2018 Feb 13. PMID 29433339
- [Background] Marechal C, Berthiller J, Tosetti S, Cogniat B, Desombres H, Bouvet L, Kassai B, Chassard D, de Queiroz Siqueira M. Children and parental anxiolysis in paediatric ambulatory surgery: a randomized controlled study comparing 0.3 mg kg-1 midazolam to tablet computer based interactive distraction. Br J Anaesth. 2017 Feb;118(2):247-253. doi: 10.1093/bja/aew436. PMID 28100529
- [Background] Kuhlmann AYR, Lahdo N, Staals LM, van Dijk M. What are the validity and reliability of the modified Yale Preoperative Anxiety Scale-Short Form in children less than 2 years old? Paediatr Anaesth. 2019 Feb;29(2):137-143. doi: 10.1111/pan.13536. Epub 2018 Dec 23. PMID 30365208
- [Background] Neville DN, Hayes KR, Ivan Y, McDowell ER, Pitetti RD. Double-blind Randomized Controlled Trial of Intranasal Dexmedetomidine Versus Intranasal Midazolam as Anxiolysis Prior to Pediatric Laceration Repair in the Emergency Department. Acad Emerg Med. 2016 Aug;23(8):910-7. doi: 10.1111/acem.12998. PMID 27129606
- [Background] Mifflin KA, Hackmann T, Chorney JM. Streamed video clips to reduce anxiety in children during inhaled induction of anesthesia. Anesth Analg. 2012 Nov;115(5):1162-7. doi: 10.1213/ANE.0b013e31824d5224. Epub 2012 Oct 9. PMID 23051880